CLINICAL TRIAL: NCT01915823
Title: Randomized, Double-Blind Trial of the Safety and Efficacy of Dymista Nasal Spray Compared to Placebo Nasal Spray in the Treatment of Children Ages >4 Years to <12 Years With Seasonal Allergic Rhinitis
Brief Title: Safety and Efficacy Trial of Dymista Nasal Spray in Children Ages 4 to 11 With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP 4008
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dymista (Active Comparator): (azelastine hydrochloride and fluticasone propionate) Nasal Spray, 137mcg/50mcg: Mode of Administration: Topical/intranasal spray
  Dose: 548 mcg azelastine hydrochloride / 200 mcg fluticasone propionate, total daily dose Regimen: 1 spray per nostril twice daily
  Interventions: Drug: azelastine hydrochloride and fluticasone propionate
- Dymista vehicle (Placebo Comparator): Dose: vehicle only Regimen: 1 spray per nostril twice daily
  Interventions: Drug: Dymista vehicle

INTERVENTIONS:
Drug: azelastine hydrochloride and fluticasone propionate
  Other Names: Dymista
  Arms: Dymista
Drug: Dymista vehicle
  Other Names: placebo
  Arms: Dymista vehicle

SUMMARY:
The purpose of this study is to determine if Dymista nasal spray is better and safer than placebo in treating children ages 4 to <12 years old who have seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages >4 years to <12 years of age, inclusive at the screening visit
* The parent/caregiver must provide written informed consent and the child must provide pediatric assent, if possible
* Willing and able to comply with the study requirements
* Have a history of seasonal allergic rhinitis (SAR) to pollen in the prevailing allergy season.
* The presence of immunoglobulin E (IgE)-mediated hypersensitivity to prevailing pollen, confirmed by a positive response to skin prick test. A histamine skin test must also be positive. A positive response for both the pollen skin test and the histamine skin test is defined as a wheal diameter of at least 4 mm larger than the negative saline control
* General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
* On the first day of the placebo lead-in period (Visit 1) subjects must have a 12-hour reflective total nasal symptoms score (rTNSS )of ≥6 and a reflective congestion score of ≥2 to qualify for entry.

At Visit 2:

* Have taken at least 6 doses of the placebo lead-in medication during the placebo lead-in period
* At Visit 2, to be eligible for entry into the double-blind treatment period, subjects must have the total of the seven lead-in symptom assessments during the past 3 days of the lead-in period including the Day of Randomization (Visit 2, Day 1):

  * a 12-hour reflective TNSS ≥ 42
  * a 12-hour reflective congestion score of ≥14

Exclusion Criteria:

* On nasal examination, the presence of any superficial or moderate nasal mucosal erosion, nasal mucosal ulceration, or nasal septum perforation (Grade 1B - 4) at either the screening visit or randomization visit
* Nasal disease(s) likely to affect deposition of intranasal medication, such as acute or chronic sinusitis, rhinitis medicamentosa, clinically significant polyposis, or clinically significant nasal structural abnormalities.
* Nasal surgery or sinus surgery within the previous year.
* The use of any investigational drug within 30 days prior to signing the informed consent/pediatric assent at Visit 1. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to azelastine hydrochloride and/or fluticasone propionate or drugs similar to azelastine hydrochloride and/or fluticasone propionate
* Respiratory tract infections within 14 days prior to Visit1
* Significant pulmonary disease including asthma. Subjects with intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
* Chronic obstructive sleep apnea syndrome (clinical diagnosis)
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug that might significantly affect the subject's ability to complete this trial
* Clinically relevant abnormal physical findings which, in the opinion of the investigator or sponsor's medical monitor, would interfere with the objectives of the study or that may preclude compliance with the study procedures
* Family members of the research center or private practice personnel who are directly involved in this study are excluded
* Members of the same household cannot be enrolled at the same time
* Subjects who have used medications or therapies that could interfere with safety and efficacy evaluations and have not had the proper washouts from these medications or therapies
* Any behavioral condition which could affect subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism
* Positive pregnancy test in female subjects ≥ 9 years of age
* Females who are pregnant or nursing
* Females of childbearing potential who are not abstinent and not practicing a medically acceptable method of contraception
* Subjects who fail to complete the symptom diary during the lead-in period, defined as missing data for >50% of entries
* Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimens following a brief period of missed injections do not preclude participation). Dose reduction when a new bottle is used does not preclude participation.
* Planned travel outside of the pollen area during the study period

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Clinical Research Center of Alabama,LLC, Birmingham, Alabama
  - Little Rock Allergy and Asthma Clinical research Center, Little Rock, Alaska
  - Clinical Research Atlanta, Atlanta, Georgia
  - Aeroallergy Research Laboratories of Savannah, Savannah, Georgia
  - Atlanta Allergy and Asthma Clinic, Stockbridge, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Clinical Research Institute of Indiana, Indianapolis, Indiana
  - Family Allergy and Asthma Reserach, Louisville, Kentucky
  - Institute for Asthma and Allergy PC, Wheaton, Maryland
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Clinical Research of the Ozarks,Inc, Warrensburg, Missouri
  - Allergy and Asthma Research NJ inc, Mount Laurel, New Jersey
  - Atlantic Research Center, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy and Asthma, Oklahoma City, Oklahoma
  - Allergy and Asthma Specialist PC, Blue Bell, Pennsylvania
  - Asthma and Allergy Research Associate, Upland, Pennsylvania
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - Allergy and Asthma Consultants, LLP, Charleston, South Carolina
  - Isis Clinical Research, LLC, Ausitn, Texas
  - Sirius Clinical Research, Austin, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Live Oak Allergy and Asthma Clinic, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Immunology/allergy and asthma Care of Waco, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Dymista: (azelastine hydrochloride and fluticasone propionate) Nasal Spray, 137mcg/50mcg: Mode of Administration: Topical/intranasal spray
  Dose: 548 mcg azelastine hydrochloride / 200 mcg fluticasone propionate, total daily dose Regimen: 1 spray per nostril twice daily
  azelastine hydrochloride and fluticasone propionate
- Dymista Vehicle: Dose: vehicle only Regimen: 1 spray per nostril twice daily
  Dymista vehicle
Period: Overall Study
Arm/Group | Dymista | Dymista Vehicle
Started | 173 | 175
Completed | 171 | 173
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dymista | Dymista Vehicle | Total
Number analyzed (Participants) | 173 | 175 | 348
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 173 | 175 | 348
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (2.11) | 8.4 (2.06) | 8.4 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 85 | 162
  Male | 96 | 90 | 186
Region of Enrollment [Number; unit: participants]
  United States | 173 | 175 | 348

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy
Description: change from baseline in AM+PM rTNSS (reflective total nasal symptoms score): ITT( intent to treat population)change from baseline in 12-hour reflective total nasal symptom score (rTNSS) consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary for the entire 14 day study period.The measurement scale is 0 to 24 so that the higher the number the worse the symptom.A reduction in symptom severity score is indicated by a negative value.A greater negative value suggests improvement.
Time Frame: 15 days of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dymista | Dymista Vehicle
Number analyzed (Participants) | 152 | 152
units on a scale | -3.83 (5.154) | -2.77 (4.731)

2. Secondary Outcome: Safety
Description: * Subject-reported adverse experiences (incidence, type, and severity of adverse events)
  * Nasal Examinations
  * Vital signs assessments
Time Frame: entire length of study (day 1 to day 22)
Measure: Number; unit: occurance
Arm/Group | Dymista | Dymista Vehicle
Number analyzed (Participants) | 173 | 175
occurance | 28 | 23

3. Other Pre Specified Outcome: Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ)
Description: Change from baseline to Visit 4 in the ITT ( intent to treat) Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) in subjects equal to or greater than 6 years old and less than12 years old compared to placebo.Scored on a 0 to 7 scale with 0 being not troubled at all and 7 being extremely troublesome. The higher the difference the better the result.
Time Frame: day 1 to day 15 of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dymista | Dymista Vehicle
Number analyzed (Participants) | 126 | 135
units on a scale | -.91 (1.22) | -.66 (1.22)

ADVERSE EVENTS:
Arm/Group | Dymista | Dymista Vehicle
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/175
Other Adverse Events (participants affected / at risk) | 13/173 | 6/175
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dymista (N=173) | Dymista Vehicle (N=175)
dysgusia (Nervous system disorders) | 7 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Meda Pharmaceuticals requests that it receive copies of any intended communication at least 15 working days for an abstract or oral presentation and 45 working days for a manuscript). This is to allow Meda Pharmaceuticals to review the communications for accuracy , to verify that confidential information is not being inadvertently divulged, to provide any relevant supplementary information, and to allow establishment of co-authorship.